CLINICAL TRIAL: NCT02237326
Title: Safety and Validity Evaluation for Cervical Cancer Screening and Treatment Techniques Among HIV-infected Women
Brief Title: Visual Inspection With Acetic Acid Compared to Lugol's Iodine in HIV-infected Women
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SSC 1825; 10-00197 (Other: University of California Committee for Human Research)
Record Dates: First submitted 2014-09-03; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; HIV
Keywords: Visual Inspection with Acetic Acid; Visual Inspection with Lugol's Iodine; Cervical Intraepithelial neoplasia; Cervical Cancer Screening; HIV infected women
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Watchful Waiting; Acetic Acid; Lugol's solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual Inspection with Lugol's Iodine (Active Comparator): Participants underwent colposcopic exam, followed by Visual Inspection with Lugol's Iodine (VILI) by a second, blinded clinician (the order of exams was reversed to eliminate potential interference with exam results due to iodine staining). Biopsy was done after the VILI.
  Interventions: Procedure: Visual Inspection with Lugol's Iodine
- Visual Inspection with Acetic Acid (Active Comparator): Participants underwent Visual Inspection with Acetic Acid followed by colposcopy by a second clinician who was blinded to the screening test result.
  Interventions: Procedure: Visual Inspection with Acetic Acid

INTERVENTIONS:
Procedure: Visual Inspection with Acetic Acid — Visual Inspection with Acetic Acid is the application of acetic acid to a cervix, followed by examination with a light source. It is not a new drug or device, and has been used in resource-limited settings for several decades. The purpose of this trial is to compare the two screening techniques, which had not been done previously.
  Arms: Visual Inspection with Acetic Acid
Procedure: Visual Inspection with Lugol's Iodine — Visual Inspection with Lugol's Iodine is the application of lugol's iodine to a woman's cervix, followed by examination with a light source with the goal of detecting precancerous lesions. Like Visual Inspection with Acetic Acid, it is not a new drug or device.
  Arms: Visual Inspection with Lugol's Iodine

SUMMARY:
The clinical trial is part of a larger study to evaluate the safety and efficacy of screening techniques for cervical cancer among HIV-infected women. The investigators randomized women to undergo screening with Visual Inspection with Acetic Acid (VIA) or Visual Inspection with Lugol's Iodine (VILI), along with a colposcopy. All outcome and treatment decisions were based on the colposcopy exam done at the study visit. The investigators then compared outcomes between the two groups to assess the test characteristics of both VIA and VILI.

DETAILED DESCRIPTION:
Cervical cancer and HIV are intersecting epidemics that both disproportionately affect low-income women; the impact of the socioeconomic disparity and biologic synergy of these two diseases is seen dramatically in Kenya, where cervical cancer is the most common cancer killer. HIV-infected women are at increased risk for the development of cervical precancer and cancer, develop more aggressive lesions and are affected at younger ages. Although screening for and treatment of precancer has reduced the incidence of cervical cancer to close to zero in resource-rich countries, strategies are costly and not available in most resource-limited countries. Novel testing and treatment methods that can be carried out in low-resource settings are urgently needed to prevent cervical cancer in these settings, especially among HIV-infected women. Using a cross-sectional study design, the investigators tested two potentially low-cost and effective cervical cancer screening methods: visual inspection with acetic acid (VIA) and protein biomarkers expressed in the presence of cervical dysplasia, neither of which have been well-studied in HIV-infected women. Investigators also randomized a small subset of women to undergo VIA compared to Visual Inspection with Lugol's Iodine (VILI) to compare the test characteristics of these two screening exams. In addition, remarkably little is known about the potential impact of the presence, diagnosis and treatment of human papillomavirus-related dysplasia on HIV genital shedding, a major risk factor for HIV transmission. To explore the impact of the presence, diagnosis and treatment of human papillomavirus-related cervical dysplasia on HIV-1 in genital secretions, investigators compared the levels of HIV-1 RNA found in the cervicovaginal secretions of women with no evidence of cervical dysplasia to levels in women with high-grade cervical dysplasia. They also compared the levels of HIV-1 RNA prior to and after cervical biopsy as well as up to 14 weeks after standard treatment for cervical dysplasia using loop electrosurgical excision procedure (LEEP). Results from this study will inform the prioritization and design of safe, effective and low-cost cervical cancer screening and prevention programs for HIV-infected

ELIGIBILITY:
Inclusion Criteria:

* 23-59
* Intact cervix/uterus
* no evidence of infection
* ability to provide informed consent

Exclusion Criteria:

* pregnant

Ages: 23 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 654 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Test Positivity Rate | eight months
  Investigators compared the test positivity between VIA and VILI.

SECONDARY OUTCOMES:
Sensitivity | 12 Months
  Investigators compared the sensitivity of VIA and VILI for the outcome of cervical intraepithelial neoplasia 2 or greater.

OTHER OUTCOMES:
Specificity | 12 months
  Investigators compared the specificity of VIA and VILI for the outcome of cervical intraepithelial neoplasia 2 or greater

CONTACTS AND LOCATIONS:
Locations (1):
- Family AIDS Care and Education Services, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Huchko MJ, Sneden J, Zakaras JM, Smith-McCune K, Sawaya G, Maloba M, Bukusi EA, Cohen CR. A randomized trial comparing the diagnostic accuracy of visual inspection with acetic acid to Visual Inspection with Lugol's Iodine for cervical cancer screening in HIV-infected women. PLoS One. 2015 Apr 7;10(4):e0118568. doi: 10.1371/journal.pone.0118568. eCollection 2015. PMID 25849627